CLINICAL TRIAL: NCT01348230
Title: Glycoproteomic Analysis of Urine in Women Undergoing Spontaneous Preterm Delivery
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1179277
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Preterm Birth
Keywords: Premature prolonged rupture of membranes; Premature labor; Uromodulin; Glycosylation
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- prior preterm delivery at 24-32 weeks: collect their first morning urine samples before each of their remaining prenatal care appointments for our studies
  Interventions: Other: Urine samples
- prior preterm delivery at 32-34 weeks: collect their first morning urine samples before each of their remaining prenatal care appointments for our studies
  Interventions: Other: Urine samples
- prior preterm delivery at 34-36 weeks: collect their first morning urine samples before each of their remaining prenatal care appointments for our studies
  Interventions: Other: Urine samples

INTERVENTIONS:
Other: Urine samples — collect their first morning urine samples before each of their remaining prenatal care appointments for our studies

SUMMARY:
When babies are premature, or born before they are fully developed, they face many different medical problems, some of which are quite devastating, such as cerebral palsy, mental retardation, blindness, deafness, severe intestinal problems, and developmental delays. Unfortunately, in more than half the cases of premature births, there is no procedure or test that an obstetrician can employ to predict if a fetus is at risk for premature birth, especially when the mother is healthy. This study seeks to determine if certain factors found in the urine undergo specific changes that can be used to detect premature births of this type before they happen.

DETAILED DESCRIPTION:
In this study, the investigators will identify women with a history of preterm delivery between 24-32 weeks, 32-34, and 34-36 weeks gestation based on diagnosis codes in the medical record who are currently pregnant. The investigators will ask these women when they are in the 16-20 week into their pregnancy to fill out a questionaire to determine study eligibility. If chosen to participate, the investigators will ask them to collect their first morning urine samples before each of their remaining prenatal care appointments for our studies. The investigators will also ask them if the investigators can check their medical records to determine if they later had a premature baby. If these women in either group give birth prematurely, then the investigators will analyze the glycoproteins in their urine samples using known values from women who did not have a premature birth as controls. If the investigators can see any changes in glycosylation in the women who gave birth prematurely, then this information will be used to apply for a larger study that will determine if such changes apply to all women. If it can then be shown to apply to all women, then the investigators may use it to predict preterm delivery. This information would allow physicians to design treatments to help these women and their babies, and spare them these disabilities. Some women go into labor prematurely, well before they should give birth. Physicians can intervene in some cases to stop labor, and allow the fetus to develop further in the mother's womb. However, in more than half the cases the physician cannot stop this process, and the baby is born prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a history of preterm delivery

Exclusion Criteria:

* Individuals that abuse alcohol or drugs
* Individuals under the age of 18
* Individuals that do not speak fluent English
* Individuals with multifetal gestation
* Individuals with known fetal anomaly
* Individuals receiving heparin treatment during current pregnancy
* Individuals with current or planned cervical cerclage
* Individuals with hypertension requiring medication
* Individuals with a seizure disorder
* Individuals who plan to deliver at some location other than the University of Missouri affiliated hospitals
* Individuals with a known abnormal fetal karyotype

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a history of preterm delivery who are currently pregnant and receiving care at affiliates of the University of Missouri, including Missouri Ob/Gyn Associates, University of Missouri Women's and Children's Hospital, and University of Missouri Center for Maternal-Fetal-Medicine and Ultrasound Clinic.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Glycosylation changes in glycoproteins in urine | After delivery of preterm infant, less than one year
  In participating women who deliver preterm, the collected urine specimens will be analyzed to evaluate glycosylation changes in glycoproteins, specifically uromodulin.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W McCullough, MD, Principal Investigator — University of Missouri Department of Obstetrics and Gynecology
Locations (1):
- University of Missouri Hospitals and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No